CLINICAL TRIAL: NCT06556537
Title: Effects of Face-to-face and Video-assisted Physical Exercise Sessions on Frailty, Mental and Physical Health of Older Adults in Rural Areas.
Brief Title: Effects of Physical Exercise on Frailty, Mental and Physical Health of Older Adults in Rural Areas.
Acronym: Rural-Frail
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Ángel Matute-Llorente, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID2022-140622OA-I00.
Record Dates: First submitted 2024-07-21; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Old Age; Frailty
Keywords: Exercise; Rural areas
MeSH Terms: conditions — Frailty; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician will only have codes but in the database but will not know which code corresponds to which group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will undergo a face-to-face and video-assisted physical exercise intervention.
  Interventions: Device: Face-to-face and video-assisted training
- Control group (No Intervention): Participants in the control group will maintain their usual lifestyle throughout the project. They will receive physical activity recommendations for older people and will attend monthly health promotion meetings.

INTERVENTIONS:
Device: Face-to-face and video-assisted training — During the first phase, the intervention group will receive face-to-face training over 12 weeks. Each session will last 60 minutes, and there will be five sessions per week, with three supervised and two unsupervised.
  In the second phase, there will be 60 work sessions, divided into blocks of four weeks on three occasions, with one month of exercise and two months of non-exercise over the remaining 9 months. This phase will be conducted via video assistance. Each session will include a warm-up of 10-15 minutes, a main part of 20-40 minutes, and a cool-down of 10-15 minutes.
  Other Names: Exercise
  Arms: Intervention group

SUMMARY:
Global aging is a significant challenge, both economically and in terms of public health. One of the main challenges is to maintain the health and functionality of older adults. Physical exercise has been suggested as one of the best non-pharmacological tools to prevent health and functionality loss. However, existing scientific literature has mainly focused on older adults from urban centers. There are no studies focused on older people in rural areas, who have particular characteristics.

The present project aims to evaluate the effects of a face-to-face and video-assisted intervention, which incorporates multi-component physical exercise with different motivational strategies, on the mental health, physical function, and frailty of individuals over 65 years of age residing in rural areas. Additionally, it aims to determine the effectiveness, safety, and adherence of new technologies in carrying out an intervention that includes multi-component physical exercise, cognitive work, and motivational strategies through video assistance for older women and men living in rural areas.

A randomized controlled trial will be conducted, involving 240 people over the age of 65 who will be randomly divided into two groups. One group, the intervention group, will participate in a face-to-face multicomponent physical exercise program three times a week for 60 minutes per session over 12 weeks. After that, the intervention will continue through video-assisted sessions for the remaining nine months, divided into three blocks of two months of rest and one video-assisted intervention. The control group will continue with their usual daily activities but receive recommendations for physical activity and mental and physical health talks. Both groups will undergo a battery of tests to evaluate the effects of the interventions. The primary variable measured will be functional capacity, assessed through the Short Physical Performance Battery. Secondary variables will include health-related physical condition (Power frail app), cognitive function (Trail making test), and quality of life, among others.

The results expected from this study will be of significant scientific and technical importance in the field of psycho-socio-health. Consequently, the project is of utmost importance, not only to enhance the health of the rural population but also to promote individual and social sustainability.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 65 years.
* Be able to provide informed consent voluntarily.
* Walk autonomously.
* Have a score of 4 points or more on the Short Physical Performance Battery (SPPB).

Exclusion Criteria:

Those that have to do with contraindications for performing physical exercise:

* Recent acute myocardial infarction within the last 3-6 months or unstable angina.
* Uncontrolled atrial or ventricular arrhythmias.
* Dissecting aortic aneurysm.
* Severe aortic stenosis.
* Acute endocarditis or pericarditis.
* Uncontrolled arterial hypertension (>180/100 mmHg).
* Acute thromboembolic disease.
* Acute and severe heart or respiratory failure.
* Recent bone fracture, orthostatic hypotension.
* Diabetes or uncontrolled hypoglycemia.
* Any pathology that causes a significant functional limitation such as advanced Parkinson's, considerable vision or hearing problems Cancer, or autoimmune disease.
* People scoring less than 4 on the SPPB (dependents).
* Any pathology or circumstance that the primary care team considers counterproductive to participation in physical exercise.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Frailty status. | T0 = pre-intervention, T1 = 3 months, T2 = 6 months, T3 = 9 months, and T4 = 12 months.
  Frailty status measured with the Short Physical Performance Battery (SPPB). The minimum value is 0 and the maximum value is 12 points. A score of < 10 points means frailty. Therefore, a higher score means a better outcome.

SECONDARY OUTCOMES:
Frailty. | T0 = pre-intervention, T1 = 3 months, T2 = 6 months, T3 = 9 months, and T4 = 12 months.
  Frailty status measured with the Frailty Trait Scale (FTS). The minimum value for the 5-item FTS is 0 and the maximum value is 50 points. Frail participants are those with FTS5 scores > 25 points. Therefore, a higher score means a worse outcome.
Power Frail App. | T0 = pre-intervention, T1 = 3 months, T2 = 6 months, T3 = 9 months, and T4 = 12 months.
  App designed to assess muscle power and frailty in older adults.
Cognitive impairment. | T0 = pre-intervention, T1 = 3 months, T2 = 6 months, T3 = 9 months, and T4 = 12 months.
  Cognitive impairment measured with the Mini Mental State Examination (MMSE) test. The minimum value is 0 and the maximum value is 30 points. Any score of 24 or more indicates a normal cognition. Therefore, higher scores indicate a worse outcome.
Mental health and depression. | T0 = pre-intervention, T1 = 3 months, and T4 = 12 months
  Mental health and depression measured with the Geriatric Depression Scale. The minimum value is 0 and the maximum value is 15 points. A score of > 5 suggests depression. Therefore, higher scores mean a worse outcome.
Quality of life of participants EuroQol-5D. | T0 = pre-intervention, T1 = 3 months, and T4 = 12 months
  Quality of life measured with the EuroQol-5D. The minimum value is 0 and the maximum value is 1. A higher score means a better outcome.
Trail Making Test (TMT). | T0 = pre-intervention, T1 = 3 months, T2 = 6 months, T3 = 9 months, and T4 = 12 months.
  Speed for attention, sequencing, mental flexibility visual search and motor function measured with the TMT parts A & B. There is no maximum value or minimum value. In the part A, a score of > 78 seconds suggests deficiency. In the part B is > 273 seconds. Results for both are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
DeJong Gierveld Loneliness Scale. | T0 = pre-intervention, T1 = 3 months, and T4 = 12 months.
  Emotional and social loneliness measured with the DeJong Gierveld Loneliness Scale. The minimum value is 0 and the maximum value is 6 points. This gives a possible range of scores from 0 to 6, which can be read as follows: 0 = (Least lonely) and 6 = (Most lonely). Therefore, higher scores mean a worse outcome.
The Aging Self-Efficacy Scale. | T0 = pre-intervention, T1 = 3 months, and T4 = 12 months.
  The perceived level of control that elderly individuals have over the aspects, content, and outcomes of aging measured with the Aging Self-Efficacy Scale. The minimum value is 10 and the maximum value is 40 points. A higher score means a better outcome.
Muscular strength of the upper limbs. | T0 = pre-intervention, T1 = 3 months, and T4 = 12 months.
  Measured with a handgrip dynamometer.
Muscular strength of the lower limbs. | T0 = pre-intervention, T1 = 3 months, and T4 = 12 months.
  Measured with the stand and sit chair test.
Aerobic capacity. | T0 = pre-intervention, T1 = 3 months, and T4 = 12 months.
  Six minute walk test.
Walking speed. | T0 = pre-intervention, T1 = 3 months, T2 = 6 months, T3 = 9 months, and T4 = 12 months.
  Walking speed measured over 3, 4, and 6 meters.
SARC-F Questionnaire. | T0 = pre-intervention, T1 = 3 months, and T4 = 12 months
  Sarcopenia measured with the SARC-F questionnaire. The minimum value is 0 and the maximum value is 10 points. A score of 4 points or more indicates a high risk of sarcopenia. Therefore, higher scores mean a worse outcome.
Body composition - Fat mass and Fat-Free mass. | T0 = pre-intervention, T1 = 3 months, and T4 = 12 months.
  Body fat measured with bioelectrical impedance analysis.
Objective physical activity levels (minutes and intensities) | T0 = pre-intervention, T1 = 3 months, and T4 = 12 months
  Physical activity levels registered with triaxial accelerometers that they will wear during 7 days.
Walking steps. | T0 = pre-intervention, T1 = 3 months, and T4 = 12 months.
  Number of walking steps measured with Global Positioning System.
Walking distance. | T0 = pre-intervention, T1 = 3 months, and T4 = 12 months
  Total walking distance, in meters, measured with Global Positioning System.
Walking speed. | T0 = pre-intervention, T1 = 3 months, and T4 = 12 months.
  Walking speed, in meters per second, measured with Global Positioning System.
Physical activity levels | T0 = pre-intervention, T1 = 3 months, T2 = 6 months, T3 = 9 months, and T4 = 12 months.
  Physical activity levels measures with Physical Activity Scale for the Elderly (PASE). It uses frequency, duration, and intensity level of activity over the previous week to assign a score, ranging from 0 to 793, with higher scores indicating greater physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Matute-Llorente, PhD, Principal Investigator — University of Zaragoza - EXERGENUD Research Group
Locations (1):
- EXERGNEUD Research Group, Zaragoza, Spain